CLINICAL TRIAL: NCT06220357
Title: Comparing Diluted to Standard Concentration Indocyanine Green Angiography: a Novel Approach to Free Flap Perfusion Evaluation in Reconstructive Microsurgery
Brief Title: Diluted Indocyanine Green Angiography: a Novel Approach to Free Flap Perfusion Evaluation in Reconstructive Microsurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Parintosa Atmodiwirjo, Medical Doctor, Indonesia University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 22-06-0636
Record Dates: First submitted 2024-01-14; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Free Flap Evaluation; Indocyanine Green Concentration; Perfusion
Keywords: Free flap; Indocyanine Green Reconstructive; Microsurgery

STUDY DESIGN:
Intervention Model Description: The population were divided into three equal groups of indocyanine green concentration : 5 mg/mL, 2,5 mg/mL, and 0,5 mg/mL
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The indocyanine green (ICG) is added into the syringe by research assistant before operation ended. Each bottle contains 25 mg of lipophilic powder with the active ingredient being ICG. It is packaged with 5 ml of sterile distilled water for dilution, resulting in a solution of 5 mg/ml. The dilution process was carried out carefully to ensure the accuracy of the concentrations. The ICG was diluted into several concentrations using sterile distilled water. The patient didn't know which concentration were given to them. The injection to the patient was performed by anesthesiologist who didn't know about the concentration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (5 mg/mL) (Experimental): This group received 5 mg/mL of ICG or 100% in terms of concentration. The 1 mL of the ICG solution was taken using a 3 mL syringe
  Interventions: Diagnostic Test: Indocyanine Green
- Group B (2,5 mg/mL) (Active Comparator): This group received 2,5 mg/mL of ICG or 50% in terms of concentration. The 0.5 mL of the ICG solution was mixed with 0.5 mL of distilled water using a 1 cc syringe
  Interventions: Diagnostic Test: Indocyanine Green
- Group C (0,5 mg/mL) (Active Comparator): This group received 0,5 mg/mL of ICG or 10% in terms of concentration. The 0.1 mL of the ICG solution was mixed with 0.9 mL of distilled water using a 1 cc syringe
  Interventions: Diagnostic Test: Indocyanine Green

INTERVENTIONS:
Diagnostic Test: Indocyanine Green — The patients were split into three different groups, the patient were given ICG with three different concentrations in a double-blind randomized manner postoperatively. The fluorescence emitted was quantitatively analyzed using the ImageJ software to ascertain the mean gray values, providing a robust measure of the ICGA concentration. The imaging was captured using a FLUORO 4000XL type NIR camera, positioned at a distance of 15-20 cm perpendicular to the flap.

SUMMARY:
The evaluation of perfusion in free flaps is crucial in clinical practice. Currently, the gold standard for evaluation is subjective through clinical assessment. However, indocyanine green angiography (ICGA), a tool that uses a near-infrared (NIR) camera to depict and monitor flap vascularization, offers an objective and reproducible alternative. The population in this study were divided into three equal groups, where each groups were assessed with Indocyanine Green (Aurogreen®, Aurolab, Tamil Nadu, India). The study was conducted with three distinct concentrations of ICGA: 5 mg/mL (100% standard concentration), 2.5 mg/mL (50%), and 0.5 mg/mL (10%). Indocyanine green was given in immediate postoperative manner, after the patient defect has been reconstructed with free flap.

DETAILED DESCRIPTION:
Indocyanine green (ICG) angiography is a novel technique for assessing tissue perfusion. The primary outcome is gray values that being evaluated with IMAGE. Through this study optimal concentration that will show fluorescence in NIR camera can be seen. This is important in order to evaluate free flap perfusion.

This study included 47 patients who underwent free flap surgery. The subjects were consisted of postoperative patient with fibular free flap (FFF), anterolateral thigh flap (ALT), radial forearm free flap (RFFF), and deep inferior epigastric perforator flap (DIEP), with inclusion criteria of this study are individuals who have successfully undergone micro-reconstruction surgery utilizing a viable free flap, with no prior surgical intervention in the area under evaluation, and the donor area for the free flap is devoid of any history of trauma or surgery.

ELIGIBILITY:
Inclusion Criteria:

* individuals who have successfully undergone micro-reconstruction surgery utilizing a viable free flap, with no prior surgical intervention in the area under evaluation, and the donor area for the free flap is devoid of any history of trauma or surgery. Furthermore, these subjects exhibit an albumin level exceeding 3 g/dL, Haemoglobin more than 10mg/dL, and no complication intraoperative

Exclusion Criteria:

* patients with a history of allergy or hypersensitivity to iodine or ICG, those with renal insufficiency or undergoing routine hemodialysis, and those regularly consuming sodium bisulfites. Additionally, patients with hepatic dysfunction, those regularly taking anticonvulsant drugs, and those experiencing complications during and post-operation are also excluded. Furthermore, patients with psychopathology and/or mental disorders, and those whose transferred free flap has experienced trauma or damage due to external factors during care are not suitable for this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Gray value of indocyanine green fluorescent | 2-5 minutes after the ICG injection
  The gray values were seen as the primary outcome to found which concentration has the best fluorescence outcome. NIR Camera, 20 cm above the flap, will assess the fluorescence due to contrast. All groups results are being evaluated with IMAGEJ to produce gray value.

CONTACTS AND LOCATIONS:
Overall Officials: Parintosa Atmodiwirjo, MD, Principal Investigator — Indonesia University
Locations (1):
- Faculty of Medicine, Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No